CLINICAL TRIAL: NCT06848439
Title: A Phase II Study of Benmelstobart Combined With Anlotinib and Chemotherapy as Neoadjuvant Therapy Followed by Surgery and Postoperative Radiotherapy in Patients With Locally Advanced Oral Cancer
Brief Title: Benmelstobart-Anlotinib-Chemo for Neoadjuvant Oral Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Collaborators: Affiliated Stomatological Hospital of Nanjing Medical University (Unknown)
Responsible Party: Principal Investigator, Lirong Wu, Chief Physician; Associate Professor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BENMEL-ANLO-CHEMO-II
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Mouth Neoplasms; Neoadjuvant Therapy; Immunotherapy; Molecular Targeted Therapy
Keywords: Mouth Neoplasms; Neoadjuvant therapy; Immunotherapy; Molecular Targeted Therapy
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benmelstobart-Anlotinib-Chemo (Experimental)
  Interventions: Drug: benmelstobart-Anlotinib-Chemo

INTERVENTIONS:
Drug: benmelstobart-Anlotinib-Chemo — Neoadjuvant Treatment Regimen :
  Benmelstobart: 1200mg, Day 1, IV (21 days per cycle); Anlotinib: 10mg, Days 1-14, orally (21 days per cycle); Cisplatin: 60mg/m², Day 1, IV (21 days per cycle); Albumin-bound Paclitaxel: 260mg/m², IV infusion, Day 1 (21 days per cycle). Total of 3 cycles.
  Surgery is performed within 2 weeks after completing neoadjuvant therapy. Postoperative adjuvant treatment is selected based on pathological grading:
  Group A (pCR): Postoperative RT alone: 40Gy/5 weeks. Group B (MPR): Postoperative RT alone: 50Gy/5 weeks. Group C (partial pathological response/no pathological response) : low and intermediate-risk patients: RT: 60Gy/6w; High-risk patients: CCRT: 60-66Gy/6-6.6w + cisplatin: 60mg/m2 Q3W, 2-3 cycles.
  All patients also received adjuvant Benmelstobart 3-4 weeks after surgery, as well as maintenance Benmelstobart for a total duration of 1 year.

SUMMARY:
Exploring the Safety and Efficacy of Benmelstobart Combined with Anlotinib and Chemotherapy as Neoadjuvant Therapy Followed by Surgery and Postoperative Radiotherapy in Patients with Locally Advanced Oral Cancer

This is a single-center, Phase II study targeting patients with stage III-IVb locally advanced oral squamous cell carcinoma who meet the inclusion and exclusion criteria. The neoadjuvant therapy consists of Benmelstobart combined with Anlotinib and chemotherapy for 3 cycles (21 days per cycle). Surgery is performed within 2 weeks after completing neoadjuvant therapy. Postoperative adjuvant treatment is selected based on pathological grading:

Group A (Pathological Complete Response, pCR): Postoperative radiotherapy (RT) alone: 40Gy/5 weeks.

Group B (Major Pathological Response, MPR): Postoperative radiotherapy (RT) alone: 50Gy/5 weeks.

Group C (Partial Pathological Response/No Pathological Response):

Low-to-intermediate risk patients (no extracapsular nodal extension and negative margins): RT: 60Gy/6 weeks.

High-risk patients (extracapsular nodal extension and/or positive margins): Concurrent chemoradiotherapy (CCRT): 60-66Gy/6-6.6 weeks + Cisplatin: 60mg/m² every 3 weeks, 2-3 cycles.

Additionally, all patients will receive adjuvant Benmelstobart 3-4 weeks after surgery, followed by Benmelstobart maintenance therapy (total treatment duration of 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must meet all of the following criteria to be eligible for inclusion in this study:
* Age 18-75 years;
* ECOG PS score of 0-1;
* Pathologically confirmed untreated oral squamous cell carcinoma patients, classified as stage III-IVb according to the AJCC (8th edition) staging system;
* Women of childbearing potential must have taken reliable contraceptive measures or have a negative pregnancy test (serum or urine) within 7 days prior to enrollment, and be willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last dose of the study drug, or be surgically sterilized. For men, they must agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last dose of the study drug, or be surgically sterilized;

Signed informed consent form by the participant, with good compliance.

Exclusion Criteria:

Potential subjects must be excluded from the study if they meet any of the following criteria:

* Prior treatment with PD-1/PD-L1/CTLA-4 antibodies.
* Tumor invasion of major blood vessels.
* Requirement for systemic corticosteroid therapy (>10 mg prednisone equivalent per day) or other immunosuppressive treatment within 14 days before administration or during treatment. Inhaled or topical steroids and adrenal corticosteroid replacement therapy at ≤10 mg/day prednisone equivalent are allowed in the absence of active autoimmune disease.
* History of any active immune-related or autoimmune disease, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Active or uncontrolled severe infection (≥ Grade 2 NCI CTCAE v5.0 infection) within 4 weeks prior to enrollment.
* Coagulation disorders (INR >1.5, prothrombin time (PT) > ULN + 4 sec, or APTT >1.5 × ULN), a tendency for bleeding, or undergoing thrombolytic or anticoagulant therapy. Note: The use of low-dose heparin (adult daily dose of 6,000-12,000 U) or low-dose aspirin (daily dose ≤100 mg) for prophylactic purposes is allowed if INR ≤1.5.
* Imaging evidence of tumor invasion of major blood vessels or tumors highly likely to invade major blood vessels and cause fatal hemorrhage during the study, as assessed by the investigator.
* Any signs or history of a bleeding tendency, regardless of severity. Patients with bleeding or hemorrhagic events (≥CTCAE Grade 2) within 4 weeks prior to randomization, or those with unhealed wounds, ulcers, or fractures.
* Major organ dysfunction:

Hematological abnormalities (without correction via blood transfusion, blood products, G-CSF, or other hematopoietic stimulants within 14 days):

1. Hemoglobin (HB) <90 g/L.
2. Absolute neutrophil count (ANC) <1.5 × 10⁹/L.
3. Platelets (PLT) <100 × 10⁹/L.

Biochemical abnormalities:

1. Total bilirubin (TBIL) >1.5 × ULN.
2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 × ULN.
3. Serum creatinine (Cr) >1.5 × ULN or creatinine clearance rate (CCr) <60 mL/min. Doppler ultrasound abnormalities: Left ventricular ejection fraction (LVEF) <60%.

Thyroid function abnormalities: TSH > ULN with abnormal T3 and T4 levels. Renal dysfunction: Urine protein ≥++ on urinalysis or confirmed 24-hour urine protein level ≥1.0 g.

* History of myocardial ischemia (≥Grade I), myocardial infarction, arrhythmia (QTc ≥480 ms), or ≥Grade 2 congestive heart failure (NYHA classification) within 6 months before enrollment.
* Diagnosis of another malignancy within 3 years prior to enrollment.
* Any severe and/or uncontrolled disease, including:

  1. Poorly controlled hypertension (systolic BP ≥150 mmHg or diastolic BP ≥100 mmHg), history of myocardial ischemia (≥Grade I), myocardial infarction, arrhythmia (QT interval ≥430 ms), or heart failure (NYHA Grade I).
  2. Active or uncontrolled severe infection.
  3. Liver cirrhosis, decompensated liver disease, or active hepatitis (HBV or HCV).
  4. Poorly controlled diabetes (fasting blood glucose (FBG) >10 mmol/L).
  5. Urine protein ≥2+ and confirmed 24-hour urine protein >1.0 g.
* Presence of long-term unhealed wounds or fractures.
* Lung hemorrhage (>Grade 1 NCI CTC AE v4.0) within 4 weeks before enrollment or hemorrhage in other areas (>Grade 2 NCI CTC AE v4.0) within 4 weeks before enrollment. Patients with a tendency to bleed (e.g., active gastrointestinal ulcers) or those receiving thrombolytic or anticoagulant therapy (e.g., warfarin, heparin, or similar agents).
* History of gastrointestinal perforation and/or fistula within 6 months before treatment initiation; or history of arterial/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism.
* Imaging evidence of tumor invasion of major blood vessels or tumors highly likely to invade major blood vessels and cause fatal hemorrhage, as assessed by the investigator.
* Clinically significant ascites, including any detectable ascites on physical examination or ascites requiring treatment. Patients with only mild asymptomatic ascites detected by imaging may be enrolled.
* Uncontrolled metabolic disorders or other non-malignant systemic diseases or conditions secondary to cancer that may pose a high medical risk and/or create uncertainty in survival assessment.
* Participation in other anti-tumor clinical trials within 4 weeks prior to enrollment.
* History of substance abuse that cannot be discontinued or the presence of psychiatric disorders.
* Any other conditions determined by the investigator that may pose serious risks to patient safety, confound study results, or affect the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival at 2 years, DFS | Two years after enrollment

SECONDARY OUTCOMES:
ORR | Ten weeks after enrollment (after completion of neoadjuvant therapy)
  Objective Response Rate (ORR) as per RECIST 1.1 Criteria
Major pathological response, MPR | Twelve weeks after enrollment (after neoadjuvant therapy and surgery)
pCR | Twelve weeks after enrollment (after neoadjuvant therapy and surgery)
  Pathological complete response (pCR) rate; It was defined as the presence of 0% viable tumor on pathological examination of the tissue specimen
LRFS at 2 years | Two years after enrollment
  Locoregional Recurrence-Free Survival (LRFS)
DMFS at 2 years | Two years after enrollment
  Distant Metastasis-Free Survival(DMFS)
OS at 2 years | Two years after enrollment
  Overall Survival(OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Stomatological Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Protecting patient privacy